CLINICAL TRIAL: NCT02854072
Title: A Prospective, Randomized, Open-label, Multicenter, Parallel Design, Phase III Study to Assess the Efficacy and Safety of GV1001 Concurrent With Gemcitabine/Capecitabine Versus Gemcitabine/Capecitabine Alone in Treating Locally Advanced and Metastatic Pancreatic Cancer Patients
Brief Title: A Phase III Study to Assess the Efficacy and Safety of GV1001-Gem/Cap vs Gem/Cap in Pancreatic Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KG 4/2015
Record Dates: First submitted 2015-08-31; First posted 2016-08-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: GV1001
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — GV1001 peptide; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GV1001 + gemcitabine/capecitabine (Experimental)
  Interventions: Drug: GV1001; Drug: Gemcitabine; Drug: Capecitabine
- gemcitabine/capecitabine (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: GV1001 — At week 1, GV1001 will be administered intradermally on day 1, day 3 and day 5. This will be followed by a once weekly schedule for weeks 2, 3, 4 and 6. After that, GV1001 will be administered once monthly until withdrawal from trial treatment due to patient choice, intolerable toxicity or disease progression. GM-CSF will be used as an adjuvant, given 10-15 minutes prior to each administration of GV1001.
  Other Names: Tertomotide
  Arms: GV1001 + gemcitabine/capecitabine
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 will be intravenously administered on day 1,8 and 15 followed by 7 days' rest.
Drug: Capecitabine — Capecitabine 830 mg/m^2 will be orally given in the morning and evening (total dose of 1660 mg/m^2) for 21 days followed by 7 days' rest.

SUMMARY:
To assess treatment of GV1001 concurrent with Gemcitabine/Capecitabine versus Gemcitabine/Capecitabine alone in locally advanced and metastatic pancreatic cancer patients.

DETAILED DESCRIPTION:
This study is designed as a phase III, prospective, randomized, open-label, multicenter clinical trial comparing GV1001 concurrent with Gemcitabine/Capecitabine versus Gemcitabine/Capecitabine alone in treating locally advanced and metastatic pancreatic cancer patients. Patients will be treated until disease progression and will be subject to follow-up until death.

Patients will be randomized equally between the two arms:

1. Gemcitabine and Capecitabine
2. GV1001+ Gemcitabine and Capecitabine

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. Histologically or cytologically proven pancreatic ductal adenocarcinoma carcinoma or undifferentiated carcinoma of the pancreas.
3. Locally advanced or metastatic disease precluding curative surgical resection or patients who have relapsed following previously resected pancreatic cancer.
4. Contrast enhanced CT scan of the thorax, abdomen and pelvis within 28 days (and up to a maximum of 32 days) prior to commencing treatment.
5. Unidimensionally measurable disease (from CT scan) in accordance with the RECIST guidelines.
6. ECOG performance status 0, 1 or 2.
7. Adequate organ function as determined by the following laboratory values:

   * Platelets ≥100 x 10^9 /L
   * WBC ≥ 3 x 10^9 /L
   * ANC ≥1.5 x 10^9 /L
   * Serum total bilirubin ≤ 2.0 mg/dL
   * CCr (Cockcroft & Gault) > 50 mL/min
8. Life expectancy ≥ 90 days
9. Fully informed written consent given.

Exclusion Criteria:

1. Brain metastasis or meningeal carcinomatosis.
2. Clinically significant serious disease or organ system disease not currently controlled on present therapy.
3. Previous chemotherapy for locally advanced and metastatic disease. Previously adjuvant chemotherapy for resected pancreatic cancer will be permitted providing chemotherapy was completed more than 12 months previously.
4. Radiotherapy within the last 8 weeks prior to start of study treatment.
5. Concurrent malignancies or invasive cancers diagnosed within the past 5 years except for adequately treated basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix or resected pancreatic cancer.
6. Medication which might affect immunocompetence e.g. chronic treatment with long term steroids or other immunosuppressant for an unrelated condition. Patients will be eligible if they have been receiving short term steroids for palliation of cancer related symptoms.
7. Administration of medicines from other clinical trials within 8 weeks from registration.
8. Pregnancy or breast feeding.
9. Uncontrolled angina pectoris.
10. Known malabsorption syndromes.
11. Patients with a known hypersensitivity to any of the investigational products or patients with a dihydropyrimidine dehydrogenase (DPD) deficiency.
12. All men or women of reproductive potential, unless using at least two contraceptive precautions, one of which must be a condom.
13. Investigator's judgment against participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | one year

SECONDARY OUTCOMES:
Time to tumor progression (TTP) | one year
Objective response rate (ORR) | one year
  Objective response rate assesses by CT scan (RECIST and irRC criteria).
Clinical benefit response (CBR) | one year
Clinical response with eotaxin level (baseline of serum eotaxin level, pg/mL) | one year
Quality of Life using EORTC QLQ-C30 | up to one year
Quality of Life using EQ-5D-3L | up to one year
Change in CA19-9 (Serum cancer antigen) over time | one year
  Cancer antigen 19-9 (CA 19-9) is used to help differentiate between cancer of the pancreas and other conditions, as well as to monitor treatment response and recurrence.
Toxicity according to the NCI CTCAE v4.03 | one year

CONTACTS AND LOCATIONS:
Overall Officials: Si Young Song, M.D., Study Chair — Severance Hospital; Yong-Tae Kim, M.D., Principal Investigator — Seoul National University Hospital; Ho Soon Choi, M.D., Principal Investigator — Hanyang University Seoul Hospital; Ho Gak Kim, M.D., Principal Investigator — Daegu Catholic University Medical Center; Hong Sik Lee, M.D., Principal Investigator — Korea University Anam Hospital; Young Woo Choi, M.D., Principal Investigator — Konyang University Hospital; Gwang Ha Kim, M.D., Principal Investigator — Pusan National University Hospital; Kwang Hyuck Lee, M.D., Principal Investigator — Samsung Medical Center; Jae Hee Cho, M.D., Principal Investigator — Gachon University Gil Medical Center; Joung-Ho Han, M.D., Principal Investigator — Chungbuk National University Hospital; Seung Ok Lee, M.D., Principal Investigator — Chonbuk National University Hospital; Chang-Hwan Park, M.D., Principal Investigator — Chonnam National University Hospital; Eun Kwang Choi, M.D., Principal Investigator — Jeju National University Hospital; Kyong Joo Lee, M.D., Principal Investigator — Wonju Severance Christian Hospital; Jae Yong Cho, M.D., Principal Investigator — Gangnam Severance Hospital; Woo Jin Lee, M.D., Principal Investigator — National Cancer Center
Locations (16):
- South Korea (16):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Pusan National University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Gangnam Severance Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jo JH, Kim YT, Choi HS, Kim HG, Lee HS, Choi YW, Kim DU, Lee KH, Kim EJ, Han JH, Lee SO, Park CH, Choi EK, Kim JW, Cho JY, Lee WJ, Moon HR, Park MS, Kim S, Song SY. Efficacy of GV1001 with gemcitabine/capecitabine in previously untreated patients with advanced pancreatic ductal adenocarcinoma having high serum eotaxin levels (KG4/2015): an open-label, randomised, Phase 3 trial. Br J Cancer. 2024 Jan;130(1):43-52. doi: 10.1038/s41416-023-02474-w. Epub 2023 Oct 30. PMID 37903909